CLINICAL TRIAL: NCT05397938
Title: A Randomized, Double-blind, Double-dummy, Positive-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of JMT103 in the Treatment of Glucocorticoid Induced Osteoporosis
Brief Title: Efficacy and Safety of JMT103 in the Treatment of Glucocorticoid Induced Osteoporosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JMT103-CSP-006
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2021-12

CONDITIONS: Glucocorticoid Induced Osteoporosis
MeSH Terms: interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JMT103 60 mg group (Experimental): Patients will be administrated with JMT103 60 mg subcutaneously every 6 months (Q6W) and alendronate sodium tablet placebo once every week (QW).
  Interventions: Drug: JMT103; Drug: Alendronate sodium placebo
- JMT103 90 mg group (Experimental): Patients will be administrated with JMT103 90 mg subcutaneously every 6 months (Q6W) and alendronate sodium tablet placebo once every week (QW).
  Interventions: Drug: JMT103; Drug: Alendronate sodium placebo
- Alendronate sodium group (Active Comparator): Patients will be administrated with alendronate sodium tablet orally 70 mg weekly (QW) and JMT103 placebo subcutaneously every 6 months (Q6W).
  Interventions: Drug: Alendronate sodium; Drug: JMT103 placebo

INTERVENTIONS:
Drug: JMT103 — JMT103, subcutaneous injection, once every 6 months (Q6M)
  Arms: JMT103 60 mg group; JMT103 90 mg group
Drug: Alendronate sodium — Alendronate sodium tablet, once every week (QW)
  Arms: Alendronate sodium group
Drug: JMT103 placebo — JMT103 placebo, subcutaneous injection, once every 6 months (Q6M)
  Arms: Alendronate sodium group
Drug: Alendronate sodium placebo — Alendronate sodium tablet placebo, once every week (QW)
  Arms: JMT103 60 mg group; JMT103 90 mg group

SUMMARY:
This is a randomized, double-blind, double-dummy, positive-controlled phase II interventional study designed to evaluate the efficacy and safety of JMT103 in the treatment of glucocorticoid induced osteoporosis patients. Patients will be enrolled and randomized to 3 treatment groups, JMT103 60 mg group (and alendronate sodium tablet placebo), JMT103 90 mg group (and alendronate sodium tablet placebo), and alendronate sodium 70 mg active comparator group (and JMT103 placebo). The primary outcome measure is percent change from baseline in lumbar bone mineral density (BMD) at 12 months of treatment. Besides, percent change of lumbar BMD at 6 months, percent change of total hip and femoral neck BMD at 12 months, and the incidence of new fracture at 12 months will be evaluated. Biomarkers of s-CTX and PINP, PK evaluation of JMT103 serum drug concentration, immunogenicity evaluation of ADA and Nab, and adverse events will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* 1. Both genders aged 18 years or above, capable of autonomous action;
* 2. In the course of an ongoing glucocorticoid treatment for at least 3months with prednisone≥7.5 mg or its equivalent taken currently, and expected to be treated of no less than 6 months in total;
* 3. Any of the followings: a. History of osteoporotic fracture; b. Age≥50 years and lumbar (L1-L4) or total hip BMD of T≤-2.0 by DXA; c. Age≥40 years and a predicted 10-year risk of major osteoporotic fractures ≥ 10% (vertebral body, forearm, hip, shoulder) or a predicted 10-year risk of hip fracture ≥ 1% estimated by hormone adjusted FRAX;
* 4. At least two lumbar vertebrae from L1 to L4 evaluable by DXA;
* 5. Uncompromised ability to maintain good communication with investigator and comply with all required study procedures;
* 6. A signed informed consent under the capability of thorough understanding.

Exclusion Criteria:

* 1. Currently pregnant or lactating; For those of child bearing potential, refusal to use effective forms of contraception from signing informed consent to 6 months after last administration;
* 2. Previous or ongoing osteomyelitis or necrosis of jaw; Unhealed dental/oral operation wound; Acute jaw bone or dental disease requiring oral surgery; Planned invasive dental surgery during the study period;
* 3. Selected into other clinical studies of which the latest administration is less than 4 weeks (or 5 elimination half-lives, whichever is longer) from the first administration in this study;
* 4. Intravenous use of bisphosphonates, fluoride or strontium in the past 5 years; Oral bisphosphonates use for more than 3 years in total, or between 3 months to 3 years in total with the last medication used in the past 1 year prior to signing informed consent;
* 5. Receptor Activator for Nuclear Factor-κ B Ligand (RANKL) antibody used within 6 months prior to screening;
* 6. Administration of any of the following bone metabolism affecting drugs within 3 months prior to screening: a. Parathyroid hormone (PTH) or PTH derivatives (e.g., teriparatide); b. Anabolic hormones or testosterone; c. Sex hormone replacement; d. Selective estrogen receptor modulators (SERMs, e.g., raloxifene); e. Calcitonin; f. Other bone metabolism activating drugs include anticonvulsants (except benzodiazepines) and heparin; g. Long-term systemic use of ketoconazole, adrenocorticotropic hormone (ACTH), cinacalcet, aluminium, lithium, protease inhibitor, methotrexate or gonadotropin releasing hormone agonist;
* 7. Administration of any of the following biologic agents within 4 weeks prior to screening: a. Anti-alpha 4 integrin antibody (e.g., natalizumab); b. Anti CD4/CD8 T-cells (e.g., alefacept); c. Anti-IL12/anti-IL23 (e.g., ustekinumab); d. CTLA4 inhibitor (e.g., abatacept); e. IL1 receptor antagonist (e.g., anakinra); f. IL6 inhibitor (e.g., tocilizumab); g. Monoclonal antibody to CD20 (e.g., rituximab); h. TNF antagonist (e.g., adalimumab, certolizumab, golimumab, etanercept, infliximab);
* 8. Requirement of >1 biologic agent (other than trial drug) for the treatment of underlying inflammatory disease;
* 9. Bone metabolic disorders (other than osteoporosis alone): a. Hypo- or hyperparathyroidism; b. Osteogenesis imperfecta; c. Malignant tumor; d. Hypopituitarism; e. Hyperprolactinemia; f. Acromegaly; g. Paget disease of bone;
* 10. Hyperthyroidism or hypothyroidism, except for a stable replacement therapy for at least 3 months turning out a normal ranged TSH or increased TSH≤10.0 μIU/mL with normal ranged FT4;
* 11. Malabsorption syndrome or various gastrointestinal diseases associated with malabsorption, such as Crohn's disease and chronic pancreatitis
* 12. Liver cirrhosis or unstable liver disease (defined as ascites, hepatic encephalopathy, coagulation disorder, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice); Known or clinically significant biliary abnormalities judged by investigator (except Gilbert syndrome, asymptomatic gallstones and gallbladder polyps);
* 13. Previous organ or bone marrow transplantation;
* 14. Unwilling to take vitamin D and calcium supplements as the procedure requires;
* 15. Uncontrolled concurrent diseases, including but not limited to: uncontrolled diabetes (> 2 grade according to NCI-CTCAE5.0), symptomatic congestive heart failure, hypertension with blood pressure greater than 150/90 mmHg after standard treatment, unstable angina pectoris, arrhythmia requiring medication or instrument treatment, myocardial infarction history within 6 months, and echocardiography with left ventricular ejection fraction < 50%;
* 16. 25[OH] vitamin D level < 20 ng/mL, retest allowed after 5000 iu/day vitamin D added for 4-6 weeks;
* 17. Current hypocalcemia or hypercalcemia, defined as albumin-corrected serum calcium level of ≤ 2.2 mmol/L (8.8 mg/dL) or ≥ 2.9 mmol/L (11.5 mg/dL) (no supplementation of calcium for at least 8 hours before test);
* 18. Serum whole parathyroid hormone (iPTH) > 65 pg/mL;
* 19. Any of the followings: a. Routine blood test (shall no treatment such as blood transfusion or hematopoietic stimulating factor was received within 7 days): absolute neutrophil count < 1.5×10^9/L, platelet < 75 × 10^9/L, or hemoglobin < 90 g/L; b. Liver function test: total bilirubin > 1.5 × upper limit of normal value (ULN), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × ULN (retest allowed after 2-4 weeks for AST and ALT); c. Renal function test: estimated glomerular filtration rate (eGFR) < 35 L/(min·1.73m^2); d. Coagulation function test: activated partial thromboplastin time > 1.5 × ULN, or international normalized ratio (INR) > 1.5 × ULN;
* 20. Active bacterial or fungal infections requiring systematic treatment within 7 days prior to randomization;
* 21. HIV infection, active hepatitis, known or suspected active tuberculosis;
* 22. Any malignant tumor within 5 years prior to screening, except those expected to be cured (e.g., completely resected in situ skin basal cell or squamous cell carcinoma, cervical cancer or breast ductal cancer, etc.);
* 23. Known allergic/hypersensitive reaction or intolerance to JMT103, positive control drug, calcium and vitamin D;
* 24. Contraindicated to alendronate therapy: abnormalities of the esophagus which delay esophageal emptying (e.g., stricture or achalasia), or inability to stand or sit upright for at least 30 minutes;
* 25. BMD measurement by DXA interrupted: < 2 measurable lumbar vertebrae; Interrupting height, weight or waist circumference; Severe scoliosis and other measurement affecting conditions;
* 26. Considered unsuitable for the research project by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change rate of lumbar bone mineral density (BMD) from baseline at 12 months | 12 months

SECONDARY OUTCOMES:
Change rate of lumbar spine BMD from baseline at 6 months | 6 months
Change rate of total hip and femoral neck BMD from baseline at 12 months | 12 months
Change rate of serum type I collagen cross-linked C-terminal peptide (s-CTX) and procollagen type I N-terminal propeptide (PINP) from baseline at 1, 3, 6 and 12 months | 1, 3, 6 and 12 months
Incidence of new fractures at 12 months (vertebral and non-vertebral) | 12 months
Types and proportions of adverse events | signing informed consent - 6 months after the last administration
JMT103 serum drug concentration | Day 1 - 12 months
Incidence of JMT103 anti-drug antibodies (ADA) and neutralizing antibodies (Nab) | Day 1 - 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China